CLINICAL TRIAL: NCT06032286
Title: Evaluation of Efficacy and Safety of the Skinstylus Sterilock Microneedling System for the Treatment of Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beauty Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASIRC_SSMS_07-14-23
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Subjects Displaying Facial Ageing
Keywords: Wrinkles; Facial ageing; Micro needling

STUDY DESIGN:
Intervention Model Description: Single group, all subjects will receive intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Microneedling (Experimental): 4 microneedling sessions at baseline and days 30, 60 and 90.
  Interventions: Device: Skinstylus microneedling device

INTERVENTIONS:
Device: Skinstylus microneedling device — Microneedling, also known as percutaneous collagen induction (PCI), is a minimally invasive technique where small needles create microscopic wounds in the skin inducing collagen formation.

SUMMARY:
To assess the efficacy and safety of the Skin stylus Sterilock microneedling system in reducing the appearance of facial wrinkles.This study is intended to be a single arm study. Suitable subjects who meet all inclusion criteria and consented will undergo 4 microneedling sessions at baseline and days 30, 60 and 90.

Subjects will be assessed at days 90, 120 and finally at day 150 by a physician utilizing the wrinkle grading scale developed by Lemperle (2001) and skin laxity and texture using a modified Alexiandes Armenakas (2010) grading scale.

DETAILED DESCRIPTION:
This study is intended to be a single arm study. Suitable subjects who meet all inclusion criteria and consented will undergo 4 microneedling sessions at baseline and days 30, 60 and 90.

Subjects will be assessed at days 90, 120 and finally at day 150 by a physician utilizing the wrinkle grading scale developed by Lemperle (2001) and skin laxity and texture using a modified Alexiandes Armenakas (2010) grading scale.

Physicians will grade treatment response on days, 90, 120 and finally on day 150 using a Global Aesthetic Improvement Scale (GAIS) Standard photography will be recorded at baseline and days 30, 60, 90, 120 and finally at day 150.

Subjects will complete diaries including self-assessment of treatment response, side effects & downtime up to 7 days post treatment.

Subjects will assess treatment response on days 90, 120 and finally on day 150 using a Subject Global Aesthetic Improvement Scale (SGAIS).

Subjects will assess treatment response and satisfaction at baseline and day 150 using the Facial Appearance, Health-Related Quality of Life and Adverse Effects (FACE-Q3) Patient reported outcome measure (PROM).

The number, type and severity of adverse events will be recorded during the duration of the study period.

At the end of the study period, photography will be assessed by three blinded physicians using the wrinkle grading scale developed by Lemperle (2001)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male & females; 35 to 75 years of age with signs of facial aging.
* Fitzpatrick I-VI phototype skin types.
* Volunteers with wrinkle grading of 1 to 4 according to Lemperle (2001) wrinkle grading scale.
* Volunteers with a laxity grading of 1-3.5 according to Alexiandes Armenakas (2010) grading scale.
* Written informed consent is given.
* Females of childbearing potential (FOCBP) and females who are premenses must be willing to practice effective contraception for the duration of the study. (Effective contraception is defined as stabilized on oral contraceptive for at least 3 months, intrauterine device, condom with spermicide, diaphragm with spermicide, implant, NuvaRing, injection, transdermal patch or abstinence.)
* Females on birth control pills must have taken the same type of pill for at least 3 months prior to entering the study and must not change type during the study.
* Those who have used birth control pills in the past must have discontinued usage at least 3 months prior to the start of the study.
* Volunteers agree NOT to use any topical agents containing active ingredients such as retinol, glycolic acid in the treatment area, during the study period.
* Volunteers agree NOT to undergo any aesthetic treatments (such as Botox, fillers, microdermabrasion, laser surfacing etc.) in the treatment area, during the study period.

Exclusion Criteria:

* Volunteers have used a topical anti-aging product containing active ingredients within 4 weeks of commencing the study.
* Volunteers suffer from Hemophilia or other clotting/bleeding disorders.
* Volunteers taking anticoagulant therapy, e.g., warfarin, heparin.
* Volunteers who have used aspirin continuously in the last 2 weeks.
* Volunteers with active acne vulgaris of the face.
* Volunteers who have stopped taking birth control pills within the last 3 months.
* Volunteers suffer from uncontrolled diabetes mellitus.
* Volunteers with known malignancy and/or undergoing chemotherapy, radiotherapy, or high doses of corticosteroids.
* Volunteers suffer from keloid scars, Human Papilloma virus (HPV) or birth marks in the treatment area.
* Volunteers have a tendency for keloid scar formation.
* Volunteers suffer from eczema or skin rashes in the treatment area.
* Volunteers suffer from systemic infections such as hepatitis.
* Volunteers have known allergy to topical/local anesthetics.
* Volunteers have continuously used high dose NSAIDs for the last 2 weeks.
* Volunteers have undergone plastic surgery in the treatment area within the last 6 months.
* Volunteers have undergone filler injections in the treatment area within the last 6 months.
* Volunteers have received Botox or other neuromodulators injections in the treatment area within the last 6 months.
* Females who are pregnant, breast-feeding or who wish to become pregnant during the study period.
* Enrolled in another clinical trial during the same study period.
* Volunteer has a planned hospital admission and/or surgical procedure for an illness or disease which existed before enrolment into the clinical trial, and which may interfere with the course or outcome of the study.
* Volunteering has medical or psychological condition(s) associated with a risk of poor protocol compliance (e.g., alcoholism or drug abuse).
* Volunteer is undergoing or is likely to undergo other treatments.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Wrinkle improvement | 120 and 150 days after the first treatment
  Mean improvement over baseline of one grade for wrinkles utilizing the Lemperle (2001) grading scale scores of the periorbital, cheek folds and glabellar lines 120 and 150 days after the first treatment.
  The Lemperle Wrinkle Grading Scale, is used to assess the severity of facial wrinkles.
  The scale divides the face into distinct facial areas (horizontal forehead lines, glabellar frown lines, periorbital lines, preauricular lines, cheek folds, nasolabial folds, upper lip lines, corner of mouth line, marionette lines and chin crease). Each area is classified 0-5, (0-No wrinkles, 5-Very deep wrinkles).
  Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001;108(6):1735-1750.

SECONDARY OUTCOMES:
Texture and laxity | 120 and 150 days after the first treatment
  Mean improvement over baseline of one grade for skin laxity and texture 120 and 150 days after the first treatment using a scale developed by Alexiandes Armenakas This is a modified texture and laxity grading scale adapted from the complete grading scale developed by Alexiandes Armenakas (2010). The scale is an 8 point descriptive scale (0-4, with 0.4 increments). Where 0 is no visible evidence of skin laxity or texture and 4 is severe skin laxity and skin roughness (texture)

OTHER OUTCOMES:
Adverse events | 150 days
  Incidence and degree of (adverse events) side effects

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ablon Skin Institute, Manhattan Beach, California
  - West Dermatology Research Center, San Diego, California

IPD SHARING:
Plan to Share IPD: No
Plan for data to be published in peer reviewed journal

REFERENCES:
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Alexiades-Armenakas M. A quantitative and comprehensive grading scale for rhytides, laxity, and photoaging. J Drugs Dermatol. 2006 Sep;5(8):808-9. No abstract available. PMID 16989197
- [Background] Pusic AL, Klassen AF, Scott AM, Cano SJ. Development and psychometric evaluation of the FACE-Q satisfaction with appearance scale: a new patient-reported outcome instrument for facial aesthetics patients. Clin Plast Surg. 2013 Apr;40(2):249-60. doi: 10.1016/j.cps.2012.12.001. PMID 23506765
- [Background] Orentreich DS, Orentreich N. Subcutaneous incisionless (subcision) surgery for the correction of depressed scars and wrinkles. Dermatol Surg. 1995 Jun;21(6):543-9. doi: 10.1111/j.1524-4725.1995.tb00259.x. PMID 7773602
- [Background] Alster TS, Graham PM. Microneedling: A Review and Practical Guide. Dermatol Surg. 2018 Mar;44(3):397-404. doi: 10.1097/DSS.0000000000001248. PMID 28796657
- [Result] Ablon G. Safety and Effectiveness of an Automated Microneedling Device in Improving the Signs of Aging Skin. J Clin Aesthet Dermatol. 2018 Aug;11(8):29-34. Epub 2018 Aug 1. PMID 30214664